CLINICAL TRIAL: NCT00204685
Title: Beatmungsdauer Und Lungenfunktion Bei Beatmeten Patienten Unter Therapie Mit Dornase Alfa - Randomisierte, Doppel-Blinde, Placebo-Kontrollierte, Multizentrische, Prospektive Klinische Studie
Brief Title: Time of Ventilation and Lung Function of Ventilated Patients Under Therapy With Dornase Alfa
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Joachim Riethmueller, Dr. med. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LUFIT
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Long Term Ventilation
MeSH Terms: interventions — dornase alfa

INTERVENTIONS:
Drug: dornase alfa

SUMMARY:
The purpose of this study is to determine whether Inhalation of Recombinant Human Deoxyribonuclease Shortens Ventilation Time in Mechanically Ventilated Adults

DETAILED DESCRIPTION:
Recombinant human deoxyribonuclease I (rhDNase, dornase alpha), administered by inhalation, is currently used as a mucolytic agent in the treatment of cystic fibrosis. This prospective, randomized, placebo-controlled, double-blind clinical study should carry out whether the therapeutic use of rhDNase can be extended to adults who are undergoing long term ventilation at the intensive care. It is hypothesized that mechanically ventilated patients show elevated concentrations of DNA in airway secretions, and that these pathological DNA levels are reduced by rhDNase. The primary clinical goal of the study is to establish wether ventilation times are shortend under inhalation of rhDNAse during the ventilation time. hDNase (verum) is compared with equal amounts of 0.9% saline solution (placebo).

ELIGIBILITY:
Inclusion Criteria:

* adult
* mechanical ventilation
* expected ventilation time 3 days or longer
* full therapy is possible
* expectet ventilation time not longer than 21 days

Exclusion Criteria:

* medicinal point of view: patient won´t survive the next 21 days
* concomitant pneumococcal disease (like tuberculosis, carcinoma)
* endotracheal bleeding
* pneumothorax with no relief (e.g. thoracic drainage)
* pregnancy
* breast feeding
* participation in another clinical trail
* mechanical ventilation since more than 48 hours
* mechanical ventilation on the basis of another reason than operation, trauma or pulmonary decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2003-08; Study Completion 2006-07

PRIMARY OUTCOMES:
Time of mechanical ventilation from beginning of the ventilation-therapy up to the end of the ventilation-therapy

SECONDARY OUTCOMES:
reduction of atelectasis / dystelectasis
improval of pulmonaryfunction
reduction of pneumonia
reduction of DNA concentrations in Airway Secretions
length of stay at the Intensive Care Unit
length of stay at the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Riethmueller, Dr. med., Study Director — University Children's Hospital Tuebingen
Locations (25):
- Germany (25):
  - University Hospital, Anaesthesiology, Tübingen, Baden-Wurttemberg
  - Charité, Universitätsmedizin Berlin, Campus Mitte, Innere Intensivstation, Berlin
  - Universität Charité, Campus Mitte, Anästhesie, Intensivstation, Berlin
  - Vivantes Klinikum Spandau, Klinik für Anästhesie, Berlin
  - Klinikum Chemnitz gGmbH, Innere Medizin, Chemnitz
  - Universitätsklinikum Erlangen Medizinische Klinik, Intensivstation I, Erlangen
  - Universitätsklinikum, Innere Medizin, Intensivstation, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf, Medizinische Intensivstation, Hamburg
  - Medizinische Hochschule Hannover, Anästhesiologie, Hanover
  - Anästhesiolog. Klinik der Ruprecht-Karls-Universität, Heidelberg
  - Universitätsklinikum des Saarlandes, Innere Medizin III, Internistische Intensivstation, Homburg / Saar
  - Klinik für Anästhesiologie u. IntensivtherapieUniversität Leipzig, Leipzig
  - Universitätsklinik Lübeck, Medizinische Klinik 1, Lübeck
  - Department of internal Medicine, Lüdenscheid
  - Universität Magdeburg, Innere Medizin,, Magdeburg
  - Gutenberg-Universität, Anästhesie-Intensivstation, Mainz
  - Johannes Gutenberg-Universität Mainz, II. Medizinische Klinik, Intensivstation, Mainz
  - Johannes-Gutenberg-Universität, Neurochirurgische Klinik, Mainz
  - Universitätsklinikum Mannheim, I. Med. Klinik, Mannheim
  - Klinikum der Philipps-Universität Marburg, Intensivstation III, Marburg
  - Klinikum der Univ. München Großhadern, Anaesthesiologische Intensivstation, München
  - Klinikum der Univ. München Großhadern, München
  - Ludwig Maximilians Universität München, Großhadern, Neurologie-Intensiv, München
  - Berufsgenossenschaftliche Klinik Tuebingen, Intensive care Unit, Tübingen
  - Intensive Care Unit of the Internal Department, Universitiy of Tuebingen, Tübingen

REFERENCES:
- [Background] Aitken ML, Burke W, McDonald G, Shak S, Montgomery AB, Smith A. Recombinant human DNase inhalation in normal subjects and patients with cystic fibrosis. A phase 1 study. JAMA. 1992 Apr 8;267(14):1947-51. PMID 1548827
- [Background] Harms HK, Matouk E, Tournier G, von der Hardt H, Weller PH, Romano L, Heijerman HG, FitzGerald MX, Richard D, Strandvik B, Kolbe J, Kraemer R, Michalsen H. Multicenter, open-label study of recombinant human DNase in cystic fibrosis patients with moderate lung disease. DNase International Study Group. Pediatr Pulmonol. 1998 Sep;26(3):155-61. doi: 10.1002/(sici)1099-0496(199809)26:33.0.co;2-k. PMID 9773909
- [Background] King M, Dasgupta B, Tomkiewicz RP, Brown NE. Rheology of cystic fibrosis sputum after in vitro treatment with hypertonic saline alone and in combination with recombinant human deoxyribonuclease I. Am J Respir Crit Care Med. 1997 Jul;156(1):173-7. doi: 10.1164/ajrccm.156.1.9512074. PMID 9230743
- [Background] Rochat T, Pastore FD, Schlegel-Haueter SE, Filthuth I, Auckenthaler R, Belli D, Suter S. Aerosolized rhDNase in cystic fibrosis: effect on leucocyte proteases in sputum. Eur Respir J. 1996 Nov;9(11):2200-6. doi: 10.1183/09031936.96.09112200. PMID 8947060
- [Background] Dasgupta B, King M. Reduction in viscoelasticity in cystic fibrosis sputum in vitro using combined treatment with nacystelyn and rhDNase. Pediatr Pulmonol. 1996 Sep;22(3):161-6. doi: 10.1002/(SICI)1099-0496(199609)22:33.0.CO;2-S. PMID 8893254
- [Background] Puchelle E, Zahm JM, de Bentzmann S, Grosskopf C, Shak S, Mougel D, Polu JM. Effects of rhDNase on purulent airway secretions in chronic bronchitis. Eur Respir J. 1996 Apr;9(4):765-9. doi: 10.1183/09031936.96.09040769. PMID 8726943
- [Background] Desai M, Weller PH, Spencer DA. Clinical benefit from nebulized human recombinant DNase in Kartagener's syndrome. Pediatr Pulmonol. 1995 Nov;20(5):307-8. doi: 10.1002/ppul.1950200509. PMID 8903903
- [Background] Touleimat BA, Conoscenti CS, Fine JM. Recombinant human DNase in management of lobar atelectasis due to retained secretions. Thorax. 1995 Dec;50(12):1319-21; discussion 1323. doi: 10.1136/thx.50.12.1319. PMID 8553310
- [Background] Wills PJ, Wodehouse T, Corkery K, Mallon K, Wilson R, Cole PJ. Short-term recombinant human DNase in bronchiectasis. Effect on clinical state and in vitro sputum transportability. Am J Respir Crit Care Med. 1996 Aug;154(2 Pt 1):413-7. doi: 10.1164/ajrccm.154.2.8756815.
- [Background] Boeuf B, Prouix F, Morneau S, Marton D, Lacroix J. Safety of endotracheal rh DNAse (Pulmozyme) for treatment of pulmonary atelectasis in mechanically ventilated children. Pediatr Pulmonol. 1998 Aug;26(2):147. doi: 10.1002/(sici)1099-0496(199808)26:23.0.co;2-1. No abstract available. PMID 9727769
- [Background] Voelker KG, Chetty KG, Mahutte CK. Resolution of recurrent atelectasis in spinal cord injury patients with administration of recombinant human DNase. Intensive Care Med. 1996 Jun;22(6):582-4. doi: 10.1007/BF01708100. PMID 8814475
- [Background] Shah PL, Scott SF, Knight RA, Marriott C, Ranasinha C, Hodson ME. In vivo effects of recombinant human DNase I on sputum in patients with cystic fibrosis. Thorax. 1996 Feb;51(2):119-25. doi: 10.1136/thx.51.2.119. PMID 8711640
- [Background] Shah PL, Hodson ME. New treatment strategies in cystic fibrosis: rhDNase. Monaldi Arch Chest Dis. 1996 Apr;51(2):125-9. PMID 8680379
- [Background] Bates RD, Nahata MC. Aerosolized dornase alpha (rhDNase) in cystic fibrosis. J Clin Pharm Ther. 1995 Dec;20(6):313-5. doi: 10.1111/j.1365-2710.1995.tb00703.x. PMID 8847368
- [Background] Reiter PD, Townsend SF, Velasquez R. Dornase alfa in premature infants with severe respiratory distress and early bronchopulmonary dysplasia. J Perinatol. 2000 Dec;20(8 Pt 1):530-4. doi: 10.1038/sj.jp.7200456. No abstract available. PMID 11190594
- [Background] Durward A, Forte V, Shemie SD. Resolution of mucus plugging and atelectasis after intratracheal rhDNase therapy in a mechanically ventilated child with refractory status asthmaticus. Crit Care Med. 2000 Feb;28(2):560-2. doi: 10.1097/00003246-200002000-00045. PMID 10708200
- [Background] Shah PL, Conway S, Scott SF, Rainisio M, Wildman M, Stableforth D, Hodson ME. A case-controlled study with dornase alfa to evaluate impact on disease progression over a 4-year period. Respiration. 2001;68(2):160-4. doi: 10.1159/000050486. PMID 11287830
- [Background] Fuchs HJ, Borowitz DS, Christiansen DH, Morris EM, Nash ML, Ramsey BW, Rosenstein BJ, Smith AL, Wohl ME. Effect of aerosolized recombinant human DNase on exacerbations of respiratory symptoms and on pulmonary function in patients with cystic fibrosis. The Pulmozyme Study Group. N Engl J Med. 1994 Sep 8;331(10):637-42. doi: 10.1056/NEJM199409083311003. PMID 7503821
- [Background] Patel A, Harrison E, Durward A, Murdoch IA. Intratracheal recombinant human deoxyribonuclease in acute life-threatening asthma refractory to conventional treatment. Br J Anaesth. 2000 Apr;84(4):505-7. doi: 10.1093/oxfordjournals.bja.a013479. PMID 10823105
- [Background] Brandt T, Breitenstein S, von der Hardt H, Tummler B. DNA concentration and length in sputum of patients with cystic fibrosis during inhalation with recombinant human DNase. Thorax. 1995 Aug;50(8):880-2. doi: 10.1136/thx.50.8.880. PMID 7570441
- [Background] Grassme H, Kirschnek S, Riethmueller J, Riehle A, von Kurthy G, Lang F, Weller M, Gulbins E. CD95/CD95 ligand interactions on epithelial cells in host defense to Pseudomonas aeruginosa. Science. 2000 Oct 20;290(5491):527-30. doi: 10.1126/science.290.5491.527. PMID 11039936
- [Background] Grassmé H, Kirschnek S, Riethmueller J, Riehle A, v Kürthy G, Lang F, Weller M, Gulbins E. Role of apoptosis in Pseudomonas aeruginosa pneumonia. Science 194, 11/2001: 1783a
- [Background] 24. Riethmueller J, Grassmé H, Ziebach R, Wessels J, Eyrich M, Stern M, Gulbins E. DNA-quantification and -qualification in sputum of CF-patients for monitoring rhDNase-therapy? Journal of Cystic Fibrosis 1. 6/2002: S110
- [Background] Cook DJ, Walter SD, Cook RJ, Griffith LE, Guyatt GH, Leasa D, Jaeschke RZ, Brun-Buisson C. Incidence of and risk factors for ventilator-associated pneumonia in critically ill patients. Ann Intern Med. 1998 Sep 15;129(6):433-40. doi: 10.7326/0003-4819-129-6-199809150-00002. PMID 9735080